CLINICAL TRIAL: NCT00000261
Title: Effects of Alcohol History on Effects of Sevoflurane and Nitrous Oxide
Brief Title: Effects of Alcohol History on Effects of Sevoflurane and Nitrous Oxide - 13
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: NIDA-08391-13; R01DA008391 (NIH); R01-08391-13
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Alcohol-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; sevoflurane; ethanol; subjective effects; healthy volunteer
MeSH Terms: conditions — Alcohol-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders | interventions — Nitrous Oxide; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (1):
- Moderate drinking adults (Experimental)
  Interventions: Drug: 30% Nitrous oxide; Other: Placebo; Drug: 0.2% sevoflurane; Drug: 0.4% sevoflurane; Drug: 0.6% sevoflurane

INTERVENTIONS:
Drug: 30% Nitrous oxide
Other: Placebo — No drug (100% oxygen)
Drug: 0.2% sevoflurane
Drug: 0.4% sevoflurane
Drug: 0.6% sevoflurane

SUMMARY:
The purpose of this study is to evaluate the effects of alcohol history on the subjective and reinforcing effects of sevoflurane and nitrous oxide in healthy volunteers. All subjects underwent psychomotor testing during 4 sessions of placebo, drug/placebo, and choice of intervention.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1997-11; Primary Completion 1998-10 (Actual); Study Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
Mood | Baseline, inhalation, recovery
Psychomotor performance | Baseline, inhalation, recovery
Choice of drug vs placebo | After placebo and drug in each session

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States